CLINICAL TRIAL: NCT03061630
Title: SAMSUNG MEDICAL CENTER
Brief Title: A Prospective Study of Neoadjuvant Chemotherapy With Gemcitabine/Platinum in Muscle-Invasive or Locally-Advanced Urothelial Carcinoma of Bladder
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Park, Se-Hoon, Samsung Medical Center, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-01-006
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Urinary Bladder
MeSH Terms: interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- gemcitabine (Experimental): cisplatin 60 mg/m2 on day 1 and gemcitabine 1000 mg/m2 on days 1, 8 and 15. On day 1
  Interventions: Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Gemcitabine — D1.8.15 : GEMCITABINE 1000MG/M2
Drug: Cisplatin — D1: CISPLATIN 60G/M2

SUMMARY:
Previously-untreated, high-risk (>T3 and/or N+) muscle-invasive bladder cancer (MIBC) cisplatin 60 mg/m2 on day 1 and gemcitabine 1000 mg/m2 on days 1, 8 and 15. On day 1

DETAILED DESCRIPTION:
Screening numbers are endowed to all patients who sign the informed consent forms. These screening numbers are used as 'Subject Identification Code" along with patient initials. Patients withdrawn from the study retain their screening number. New patients must always be allotted with a new screening number. The study population includes chemotherapy-naïve adults with high-risk MIBC. Patients who meet all of the inclusion criteria and none of the exclusion criteria will receive cisplatin 60 mg/m2 on day 1 and gemcitabine 1000 mg/m2 on days 1, 8 and 15. On day 1, adequate hydration and antiemetics are needed. Study chemotherapy will repeat every 4 weeks on an outpatient basis and continued until disease progression, unacceptable toxicity, deterioration of clinical condition, patient refusal, or up to 2 or 3 cycles, depending on the operation schedules.

Patients will be seen every 4 weeks. All study subjects will be also eligible to receive best supportive care (BSC) defined as any standard supportive measures that are not considered a primary treatment of the disease under study, including the use of growth factors (i.e. G-CSF) for myelosuppression, bisphosphonates for management of skeletal metastases, analgesics and transfusion of blood products. BSC will be provided at the discretion of the investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Must be aged 20 years or more
2. Must have histologically or cytologically proven UC of bladder.
3. Must have histological evidence of high-risk muscle-invasive disease (i.e., T2~ T4) or clinically N+ disease. They must be considered to have no other treatment options than radical cystectomy.
4. Must have an ECOG performance status of 0 to 1
5. Must have a life expectancy of 6 months or more
6. At least 2 weeks since the last surgical procedures or biopsies prior to enrolment. Subjects must have recovered to <Grade 2 from all acute toxicities or toxicity must be deemed irreversible by the investigator.
7. Adequate marrow function without growth factor support or transfusion dependency
8. Adequate renal function with serum creatinine 1.5 x ULN or a calculated creatinine clearance ≥ 60 mL/min using the Cockcroft-Gault or MDRD formulas
9. Adequate hepatic function
10. Must agree to use an adequate method of contraception if the patient is sexually active, during and for 12 weeks after the completion of chemotherapy
11. Written and voluntary informed consent understood, signed and dated.

Exclusion Criteria:

1. Ongoing treatment with an anticancer agent not contemplated in this protocol
2. Radiologic finding consistent with metastatic disease
3. Severe medical or phychological illness that preclude participation to study, including any history of clinically relevant coronary artery disease or myocardial infarction within the last 3 years, (NYHA) grade III or greater congestive heart failure, cerebrovascular attack within the prior year, or current serious cardiac arrhythmia requiring medication except atrial fibrillation
4. Non-tolerable > Grade 2 neuropathy or evidence of unstable neurological symptoms within 4 weeks of Cycle 1 Day 1
5. Major surgery, other than diagnostic surgery or transurethral resection, within 4 weeks prior to Cycle 1 Day 1, without complete recovery
6. Double primary cancer of other site(s) or a history of other malignancies, except for cured ones at the discretion of investigator
7. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
8. Subjects who have exhibited allergic reactions to study treatment
9. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this study
10. Subject with legal incapacity or limited legal capacity. Dementia or significantly altered mental status that would limit the understanding or rendering of informed consent and compliance with the requirements of this protocol. Unwillingness or inability to comply with the study protocol for any reason.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
pathologic response | 30 months
  to determine the antitumor activity of study treatment in terms of pathologic response

SECONDARY OUTCOMES:
progression-free survival | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: SEHOON PARK, MD,PhD, Principal Investigator — SamsungMedicalCenter
Locations (1):
- Samsung Medical Center, Seoul, South Korea